CLINICAL TRIAL: NCT01910662
Title: Characterisation of the T-cell Response in Delayed Type Hypersensitivity Reactions to Keyhole Limpet Hemocyanin (KLH) and Tuberculin Purified Protein Derivative (PPD) in Healthy Volunteers
Brief Title: Characterisation of T-cell Response to Keyhole Limpet Hemocyanin (KLH) and Tuberculin Purified Protein Derivative (PPD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 117249
Record Dates: First submitted 2013-02-14; First posted 2013-07-29 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Dermatitis
Keywords: Suction Skin Blister; Induration; Tuberculin Purified Protein Derivative; Erythema; Biopsy; Keyhole Limpet Hemocyanin; Delayed Type Hypersensitivity
MeSH Terms: conditions — Dermatitis; Erythema; Hypersensitivity, Delayed | interventions — keyhole-limpet hemocyanin; Tuberculin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part A: (Experimental): Subjects in the Part A will receive an ID injection of 0.1 mg KLH as 0.1 mL of KLH (1 mg/mL) in the upper right forearm and an ID injection of 0.1 mL of buffer in the lower right forearm and lower and upper left forearm on Day 1.
  Interventions: Other: KLH 0.1 mg; Other: PBS (0.1 mL)
- Part B:Cohort 1A (Experimental): Subjects in the Part B Cohort 1A arm will receive a SC immunisation of 5 mg KLH in the right deltoid. On Day 15 subjects will return to the unit for an ID injection of 0.1 mg KLH as 0.1 mL of KLH (1 mg/mL) in the lower right and lower left forearm. On Day 43, 0.1mL of KLH (1 mg/mL) will be injected ID into the upper left forearm and the upper right forearm (The dose can be changed to either 5mg/1mg or 1mg/0.1mg depending on the results from the first 3 subjects in Cohort 1).
  Interventions: Other: KLH 0.1 mg; Other: KLH 5 mg
- Part B:Cohort 1B (Experimental): Subjects in the Part B Cohort 1B arm will receive a SC immunisation of 5 mg KLH in the right deltoid on Day 1. On Day 15 subjects will return to the unit for an ID injection of 0.1 mg KLH in the lower right and lower left forearm. On Day 43 subjects will then receive an ID injection of 0.1 mg KLH in the upper right and upper left forearms (The dose can be changed to either 5mg/1mg or 1mg/0.1mg depending on the results from the first 3 subjects in Cohort 1).
  Interventions: Other: KLH 0.1 mg; Other: KLH 5 mg
- Part B:Cohort 2 (Experimental): Subjects in the Part B Cohort 2 will receive an ID injection of 2TU (0.04 microg/mL) PPD in the upper right and upper left forearms on Day 1. On Day 3 (48 hours post challenge) If the induration is less than 6 mm, the subject will be re-challenged with 10 TU (0.04 microg/mL) PPD at a site at least 4 cm away from another challenge site. On Day 29 the subjects will have 2 ID injections of 2 TU or 10 TU (the same dose that produced an induration of 6 mm or more).
  Interventions: Other: Tuberculin PPD
- Part C: Cohort 1 (Experimental): Subjects in the Part C Cohort 1 will receive an ID injection of 0.1 mL PBS in the upper right forearm on Day 1. On Day 2 subjects will receive an ID injection of 0.1 ml PBS in the upper left forearm.
  Interventions: Other: PBS (0.1 mL)
- Part C: Cohort 2 (Experimental): Subjects in the Part C Cohort 2 will receive an ID injection of 2TU (0.04 microg/mL) PPD in the upper left forearms on Day 1. On Day 3 (48 hours post challenge) If the induration is less than 6 mm, the subject will be re-challenged with 10 TU (0.04 microg/mL) PPD at a site at least 4 cm away from another challenge site. On Day 29 the subjects will have 1 ID injections of 2 TU or 10 TU (the same dose that produced an induration of 6 mm or more).
  Interventions: Other: Tuberculin PPD

INTERVENTIONS:
Other: KLH 0.1 mg — KLH will be administered as single ID injection of 0.1 mg as 0.1mL of KLH (1 mg/mL)
  Arms: Part A:; Part B:Cohort 1A; Part B:Cohort 1B
Other: KLH 5 mg — KLH will be administered as single SC injection of 5 mg
  Arms: Part B:Cohort 1A; Part B:Cohort 1B
Other: PBS (0.1 mL) — PBS will be administered in Part A on Day 1 as 3 ID injections and in Part C: Cohort 1 on Day 1 and Day 2 as a single ID injection
  Arms: Part A:; Part C: Cohort 1
Other: Tuberculin PPD — Tuberculin PPD will be administered in Part B Cohort 2 on Day 1 as single ID injection of 2TU (0.04 microg/mL) in each forearm. In Part C Cohort 2 PPD will be administered on Day 1 as a single ID injection of 2TU. On day 3, if the induration is 6 mm or more; 2 ID injections of 2 TU will be administered on Day 29 in Part B Cohort 2 and 1injection of 2TU on Day 29 in Part C Cohort 2. On day 3, if the induration is less than 6 mm, subject will be re-challenged with 10 TU (0.04 microg/mL) PPD followed by 2 ID injections of 10 TU on Day 29 in Part B Cohort 2 or 1 ID injection of 10TU on Day 29 in Part C Cohort 2.
  Arms: Part B:Cohort 2; Part C: Cohort 2

SUMMARY:
This is an exploratory study to develop methodologies for the assessment of T-cell mediated therapies via skin immune challenges studies in healthy volunteers. The study will investigate what is the most appropriate; skin challenge agent, time and methodology to sample and characterise T-cells in the delayed type hypersensitivity (DTH) skin reaction. The skin challenge agents to be used in this study will be the neoantigen Keyhole Limpet Hemocyanin (KLH) and recall antigen Tuberculin Purified Protein Derivative (PPD). Part A of the study will assess an intradermal (ID) KLH challenge in three subjects to assess if the immune response to KLH is initiated by the innate or adaptive immune system. Each subject will receive one ID dose of 0.1 milligram (mg) KLH and will be assessed for a skin inflammatory response. Part B of the study will assess repeat ID challenges 28 days apart; the objective will be to characterise the T-cell response to each challenge and the kinetics of that response.

For Cohorts 1A and 1B, 16 subjects will receive an initial subcutaneous (SC) 5 mg dose of KLH. Fifteen days later the subjects will receive 0.1 mg ID KLH dose and the response will then be assessed 48 and 120 hours after the initial challenge. The ID KLH challenge will then be repeated 28 days later and the response will be assessed at 48 hours (Cohort 1A, 8 subjects) and at 120 hours (Cohort 1B, 8 subjects) post challenge. For Cohort 2, a repeat challenge of either 2 tuberculin Unit (TU) or 10 TU ID PPD will be administered 28 days apart, to 8 subjects. The first challenge response will be assessed 48 and 120 hours post challenge. The second challenge will be administered 28 days after the first and will be assessed at the same timepoints. The repeat challenge 28 days later will allow an intra-subject analysis and will determine if a subject can be used as their own control. Part C of the study will assess repeat ID challenges of PPD and PBS; the objective will be to characterise the T-cell response to each challenge and the kinetics of that response. For Cohort 1, 6 subjects will receive a 0.1ml ID dose of PBS and another dose 24 hours later. Each challenge will be assessed 48 hours post challenge. Approximately 2 subjects will have an assessment of their normal skin as a control. For Cohort 2, a repeat challenge of either 2TU or 10TU ID PPD will be administered 28 days apart, to 6 subjects. The first challenge response will be assessed 48 post challenge. The second challenge will be administered 28 days after the 1st and will be assessed at the same timepoint. The repeat challenge 28 days later will allow an intra-subject analysis and will determine if a subject can be used as their own control.

The total duration of this study for Part A is 14-18 days plus up to 30 days screening. The total duration of this study for Cohort 1A is 56-60 days plus up to 30 days screening. The total duration of this study for Cohort 1B is 59-63 days plus up to 30 days screening. The total duration of this study for Cohort 2 if 2TU is used is 45-49 days plus up to 30 day screening. The total duration of this study for Cohort 2 if 10TU is used is 48-51 days plus up to 30 days screening. The total duration of this study for Part C Cohort 1 is 15-19 days plus up to 30 day screening. The total duration of this study for Cohort 2 if 2TU is used is 42-46 days plus up to 30 day screening. The total duration of this study for Cohort 2 if 10TU is used is 45-49 days plus up to 30 days screening.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical Evaluation.
* Body weight >= 50 kg and body mass index (BMI) within the range 19.5 to 29.9 kilogram/meter squared (inclusive).
* Female subjects of non-child bearing potential. Females of child bearing potential are eligible to enter if they are not pregnant and willing to use protocol-specified methods of contraception to prevent pregnancy.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods from the time of the first dose of challenge agent until follow-up.
* Capable of giving written informed consent.
* Alanine aminotransferase (ALT) alkaline phosphatase and bilirubin <or=1.5x upper limit of normal (ULN).
* Normal electrocardiogram (ECG) measurements. Average QT duration corrected for heart rate by Fridericia's formula (QTcF) <450 millisecond (msec).
* Part B and C cohort 2 only: Subjects with a history of Bacillus Calmette Guérin (BCG) vaccination as evidence by either a BCG scar and verbal confirmation of BCG vaccination or documented medical history of a BCG vaccination with or without a BCG scar

Exclusion Criteria:

* Prior medical history of anaphylaxis, severe adverse reaction to vaccines, allergy to shellfish, asthma (excluding childhood asthma), allergic rhinitis or atopic dermatitis, severe adverse reaction to local anaesthetic, previous tuberculosis infection.
* Current treatment with beta-blockers or angiotensin converting enzyme (ACE) inhibitors.
* History of sensitivity to any of the study challenge agents or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline (GSK) Medical Monitor, contraindicates their participation.
* Received live, attenuated or recombinant vaccine(s) within 2 months of the first KLH or PPD injection or will require vaccination prior to the follow-up visit.
* Part B and C cohort 2 only: From a high risk area of the world for tuberculosis or have close family members with confirmed Mycobacterium tuberculosis (MTB).
* Antibiotics or antiviral therapy after a serious illness within 30 days of study entry.
* Immunodeficiency or autoimmunity, assessed by medical history.
* Presence of tattoos, naevi or other skin abnormalities such as keloids (or history of keloids) that may, in the opinion of the investigator, interfere with study assessments.
* Use of nicotine patches on the arm at screening that would interfere with the injection sites.
* Subjects participating, within 7 days of screening, in recreational sun-bathing, or use of sun-bed, on the area of the skin from wrist to shoulder inclusive.
* The subject has a phobia to needles or minor surgical procedures.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study.
* Use of prescription drugs or non-prescription drugs, including NSAIDs, if in the opinion of the Investigator the medication will interfere with the study procedures or compromise subject safety. Subjects must not currently take any of the following: topical steroid cream on the arms, oral or systemic steroids or any other immune-modulators.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Pregnant or lactating females.
* Donation of more than 500 milliliter (mL) blood within a 56 day period.
* Participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Part A and part B Cohort 1: The subject has received KLH SC or ID in the past.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-02-22 (Actual); Primary Completion 2013-11-26 (Actual); Study Completion 2013-11-26 (Actual)

PRIMARY OUTCOMES:
Part A: Skin inflammatory response measurement as induration by the ball point pen technique | Over a four day period after challenge
  The induration of wheals (defined as elevation and induration that are palpable in the skin) that develop as a result of intradermal immunisation with KLH or PPD will be measured in the vertical and horizontal plane using the ball point pen technique. The diameter of the induration will be measured by rolling a medium ball point pen from 10 to 20 millimetre (mm) outside the edge of the induration and toward the centre with just enough pressure to indent the skin slightly.
Part A: Skin inflammatory response measurement as erythema diameter by Laser Doppler Imaging (LDI) and ruler measurement | Over a four day period after challenge
  A Laser Doppler Imager will measure the area occupied by a given wheal and associated erythema, which reflects superficial blood flow of a subject's arm. Erythema at the immunisation site will be measured in the vertical and horizontal plane using a plastic flexible mm ruler. Measurements will be taken for both challenge agent and buffer control injections. Place the zero line of the ruler just inside the left edge of the area of erythema and read the ruler line just inside the right edge.
Part A: Skin inflammatory response measurement as induration by characterisation and measurement of the T-cells in skin biopsies | Over a three day period after challenge
  T-cells will be analysed by immunocytochemistry or other techniques to characterise the T-cells
Part B: Characterisation of T-cells in a skin DTH response | Cohort 1: Over a five day period after first challenge. Cohort 2: Over a five day period after first challenge
  Lymphocyte Activation Gene 3 (LAG 3+) T-cells collected by Punch Biopsy or skin blister will be characterised and measured by Fluorescence activated cell sorter (FACS) analysis or other immunologic techniques
Part C: Characterisation of T-cells in a skin DTH response | Cohort 1: Over a five day period after first challenge. Cohort 2: Over a three day period after first challenge
  Lymphocyte Activation Gene 3 (LAG 3+) T-cells collected by skin blister will be characterised and measured by Fluorescence activated cell sorter (FACS) analysis or other immunologic techniques

SECONDARY OUTCOMES:
Part A: Characterisation and measurement of the T-cells in skin biopsies. | At 48hrs (Day 3) after challenge
  T-cells will be analysed by immunocytochemistry or other techniques to characterise the T-cells
Part B: Skin inflammatory response measurement in Cohort 1 by the ball point pen technique | Cohort 1A: At 48hrs (Day 17) and 120hrs (Day 20) after first challenge. At Day 44 and 48hrs (Day 45) after second challenge. Cohort 1B: At 48hrs (Day 17) and 120hrs (Day 20) after first challenge. At Day 44, 45 and 120hrs (Day 48) after second challenge
  The induration of wheals (defined as elevation and induration that are palpable in the skin) that develop as a result of intradermal immunisation with KLH or PPD will be measured in the vertical and horizontal plane using the ball point pen technique. The diameter of the induration will be measured by rolling a medium ball point pen from 10 to 20 mm outside the edge of the induration and toward the centre with just enough pressure to indent the skin slightly.
Part B: Skin inflammatory response measurement in Cohort 2 by the ball point pen technique | Cohort 2: At 48hrs (Day3) and 120hrs (Day 6) after first challenge. At 48hrs (Day 31) and 120hrs (Day 34) after second challenge.
  The induration of wheals (defined as elevation and induration that are palpable in the skin) that develop as a result of intradermal immunisation with KLH or PPD will be measured in the vertical and horizontal plane using the ball point pen technique. The diameter of the induration will be measured by rolling a medium ball point pen from 10 to 20 mm outside the edge of the induration and toward the centre with just enough pressure to indent the skin slightly.
Part B: Erythema diameter measured in Cohort 1 by Laser Doppler Imaging (LDI) and ruler measurement. | Cohort 1A: At 48hrs (Day 17) and 120hrs (Day 20) after first challenge. At Day 44 and 48hrs (Day 45) after second challenge. Cohort 1B: At 48hrs (Day 17) and 120hrs (Day 20) after first challenge. At Day 44, 45 and 120hrs (Day 48) after second challenge
  A Laser Doppler Imager will measure the area occupied by a given wheal and associated erythema, which reflects superficial blood flow of a subject's arm.
Part B: Erythema diameter measured in Cohort 2 by Laser Doppler Imaging (LDI) and ruler measurement. | Cohort 2: At 48hrs (Day3) and 120hrs (Day 6) after first challenge. At 48hrs (Day 31) and 120hrs (Day 34) after second challenge.
  A Laser Doppler Imager will measure the area occupied by a given wheal and associated erythema, which reflects superficial blood flow of a subject's arm.
Part B: Characterisation and measurement of the T-cells in skin biopsies in Cohort 1. | Cohort 1A: At 48hrs (Day 17) and 120hrs (Day 20) after first challenge. At 48hrs (Day 45) after second challenge. Cohort 1B: At 48hrs (Day 17) and 120hrs (Day 20) after first challenge. At 120hrs (Day 48) after second challenge.
  T-cells will be analysed by immunocytochemistry or other techniques to characterise the T-cells
Part B: Characterisation and measurement of the T-cells in skin biopsies in Cohort 2. | Cohort 2: At 48hrs (Day3) and 120hrs (Day 6) after first challenge. At 48hrs (Day 31) and 120hrs (Day 34) after second challenge.
  T-cells will be analysed by immunocytochemistry or other techniques to characterise the T-cells
Part A and B: Number of subjects with adverse events as a measure of safety and tolerability | Part A: Day 1 to Day 4, Part B: Cohort 1A: Day 1 to Day 46.Part B: Cohort 1B:Day 1 to Day 49.Part B Cohort 2: Day 1 to 35.
  The safety and tolerability of skin challenges with KLH and PPD.administration will be assessed by adverse events (AEs), serious AE (SAE) or withdrawals due to toxicities
Part A and B: changes in clinical laboratory measurements to access safety and tolerability | Screening and up to 14 days post last visit
Part A and B: Trends in and change from baseline for blood pressure measurements | Screening and up to 14 days post last visit
Trends in and change from baseline in measure of 12-lead ECG to access safety and tolerability | Screening and up to 14 days post last visit
  Electrocardiograph (ECG) is a machine that measures the electrical activity of the heart and records changes in the hearts' rhythm.
Immediate local hypersensitivity assessment | 15-30 minutes after each SC and ID challenge immunization in each Study part/Cohort
  Examination of injection site for evidence of immediate local hypersensitivity/wheal (erythema or induration will not be taken into consideration). The diameter of the wheal (central swelling/raised skin) at immunisation site, if present at time of hypersensitivity assessment, will be measured in vertical and horizontal plane using a millimetre (mm) ruler. The average will be the diameter value. If wheal is more than 5 mm in diameter than original bleb, then subject will be labelled as having immediate local hypersensitivity (ILH) and will undergo both serum total IgE and KLH or PPD prick tes
Part A and B: Trends in and change from baseline for heart rate measurements | Screening and up to 14 days post last visit
Part C: Skin inflammatory response measurement in Cohort 2 by the ball point pen technique. | Cohort 2: At 48hrs (Day3) and 744hrs (Day 31).
  The induration of wheals (defined as elevation and induration that are palpable in the skin) that develop as a result of intradermal immunisation with PPD will be measured in the vertical and horizontal plane using the ball point pen technique. The diameter of the induration will be measured by rolling a medium ball point pen from 10 to 20 mm outside the edge of the induration and toward the centre with just enough pressure to indent the skin slightly.
Part C: Erythema diameter measured in Cohort 2 by Laser Doppler Imaging (LDI) and ruler measurement. | Cohort 2: At pre-challenge (Day1) and 48hrs (Day 3) after first challenge. At pre-challenge (Day 29) and 48hrs (Day 31) after second challenge.
  A Laser Doppler Imager will measure the area occupied by a given wheal and associated erythema, which reflects superficial blood flow of a subject's arm.
Part C: Characterisation and measurement of the T-cells in skin blisters in Cohort 2. | Cohort 2: At 48hrs (Day3) and 72hrs (Day 4) after first challenge. At 48hrs (Day 31) and 69hrs (Day 32) after second challenge.
  T-cells will be analysed by immunocytochemistry or other techniques to characterise the T-cells
Part A , B and C: Number of subjects with adverse events as a measure of safety and tolerability | Part A: Day 1 to Day 4, Part B: Cohort 1A: Day 1 to Day 46.Part B: Cohort 1B:Day 1 to Day 49.Part B Cohort 2: Day 1 to 35. Part C: Cohort 1:Day 1 to Day 19. Part C Cohort 2: Day 1 to 46.
  The safety and tolerability of skin challenges with KLH and PPD .administration will be assessed by adverse events (AEs), serious AE (SAE) or withdrawals due to toxicities
Part A, B and C: changes in clinical laboratory measurements to access safety and tolerability | Part A and B: Screening and up to 14 days post last visit. Part C: Screening and up to 14 days post last blister draw.
Part A and B: Screening and up to 14 days post last visit. Part C: Screening and up to 14 days post last blister draw. | Part A and B: Screening and up to 14 days post last visit. Part C: Screening and up to 14 days post last blister draw.
Trends in and change from baseline in measure of 12-lead ECG to access safety and tolerability | Part A and B: Screening and up to 14 days post last visit. Part C: Screening and up to 14 days post last blister draw.
  Electrocardiograph (ECG) is a machine that measures the electrical activity of the heart and records changes in the hearts' rhythm.
Immediate local hypersensitivity assessments | Part A and B: 15-30 minutes after each SC and ID challenge immunization in each Study part/Cohort. Part C: Screening and up to 14 days post last blister draw.
  Examination of injection site for evidence of immediate local hypersensitivity/wheal (erythema or induration will not be taken into consideration). The diameter of the wheal (central swelling/raised skin) at immunisation site, if present at time of hypersensitivity assessment, will be measured in vertical and horizontal plane using a millimetre (mm) ruler. The average will be the diameter value. If wheal is more than 5 mm in diameter than original bleb, then subject will be labelled as having immediate local hypersensitivity (ILH) and will undergo both serum total IgE and KLH or PPD prick tes
Part A and B: Trends in and change from baseline for heart rate measurement | Part A and B: Screening and up to 14 days post last visit. Part C: Screening and up to 14 days post last blister draw.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

REFERENCES:
- See also: Results for study 117249 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/117249?search=study&search_terms=117249#rs